CLINICAL TRIAL: NCT05311826
Title: Effectiveness of Postoperative Respiratory Physiotherapy for Pain Management in Patients Undergoing Spinal Fusion for Adolescent Idiopathic Scoliosis: a Randomized Controlled Study
Brief Title: Diaphragmatic Breathing Exercise for Patients Undergoing Arthrodesis Surgery for Adolescent Idiopathic Scoliosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RachideResp
Record Dates: First submitted 2022-03-26; First posted 2022-04-05 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2024-06

CONDITIONS: Adolescent Idiopathic Scoliosis; Spinal Fusion; Pain Management; Exercise
Keywords: spinal fusion; early rehabilitation; diaphragmatic breathing exercise; Adolescent Idiopathic Scoliosis
MeSH Terms: conditions — Agnosia; Motor Activity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: it will be masking also data analyzer
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STANDARD PHYSIOTHERAPY TREATMENT - CTL GROUP (Active Comparator): Patients aged from 12 to 24 years hospitalized for corrective arthrodesis surgery with Adolescent Idiopathic Scoliosis (AIS) diagnosis.
  Interventions: Procedure: STANDARD PHYSIOTHERAPY TREATMENT
- EXPERIMENTAL diaphragmatic breathing exercise - EXP GROUP (Experimental): Patients aged from 12 to 24 years hospitalized for corrective arthrodesis surgery with Adolescent Idiopathic Scoliosis (AIS) diagnosis.
  Interventions: Procedure: EXPERIMENTAL diaphragmatic breathing exercise

INTERVENTIONS:
Procedure: STANDARD PHYSIOTHERAPY TREATMENT — The standard postoperative rehabilitation process starts from the first postoperative day. Two sessions are provided daily, with the exception of Sunday and Saturday afternoon. A single physiotherapy session, lasting 30 minutes, can include bed exercises for upper and lower limbs and recovery of autonomy (sitting position, standing and ambulation). In this phase, the sessions are characterized by educational and counseling activities.
  The patient will be encouraged to carry out the activities independently.
  Arms: STANDARD PHYSIOTHERAPY TREATMENT - CTL GROUP
Procedure: EXPERIMENTAL diaphragmatic breathing exercise — The subjects in the intervention group (EXP) will receive, in addition to standard physiotherapy treatment, diaphragmatic breathing exercise. Four exercises in different position (supine and side lying) will be provided for each physiotherapy session by a senior physiotherapist. Patients will be instructed to perform the same exercises independently to achieve relaxation and relief of pain symptoms.
  Arms: EXPERIMENTAL diaphragmatic breathing exercise - EXP GROUP

SUMMARY:
After spinal surgery, diaphragmatic breathing exercise can be a low-cost and extremely safe intervention that can be introduced for pain management.

The aim of the study is to investigate the effectiveness of diaphragmatic breathing exercise in the management of pain in the postoperative care in patients undergoing spinal fusion for adolescent idiopathic scoliosis.

DETAILED DESCRIPTION:
Adolescent idiopathic scoliosis (AIS) is a common orthopedic condition with a prevalence of 2-3% in children aged from 10 to 16 years. It is a developmental deformity that affects both physical and psychological domains, interfering with self-esteem and mental well-being. Diagnosis is made within the first 18 years of life; in some cases, instrumented arthrodesis surgery is required, performed within the age of 25. Corrective surgery for scoliosis can be a stressful intervention for patients and their caregivers.

Postoperative pain is the major concern for patients undergoing orthopedic surgery. Significant postoperative pain also adversely affects other outcomes by hindering the healing process and delaying rehabilitation with loss of movement and walking. After arthrodesis the pain reported by the patients is significant.

Various strategies have been explored for acute pain management in patients undergoing surgery for scoliosis, with a focus on the first days post surgery. The link between breathing, lumbar spine function and pain perception is an aspect that has always been studied. The diaphragm plays an important role in spinal control and in the management of pain perception. Dysfunction of the diaphragm can lead to alterations in the biomechanics of the lumbar spine, with less proprioceptive abilities, less spinal mobility and reduced the spinal column's functionality of the tissues. Diaphragmatic rehabilitation techniques produce significant and clinically relevant improvements in the treatment of pathologies of the spine and especially in the management of painful symptoms.

A systematic review highlights how pain is able to influence the flow, frequency and volume of the respiratory act. At the same time, a regulation of breathing can be an useful tool in the control of painful symptoms.

After spinal surgery, diaphragmatic breathing exercise can be a low-cost and extremely safe tool that can be introduced for the control of painful symptoms.

The aim of the study is to investigate the effectiveness of diaphragmatic breathing exercise in the management of pain in the postoperative phase in patients undergoing arthrodesis surgery for adolescent idiopathic scoliosis.

ELIGIBILITY:
Inclusion Criteria:

* All subjects hospitalized for corrective arthrodesis surgery with Adolescent Idiopathic Scoliosis (AIS) diagnosis, aged from 12 and 24 years will be consecutively enrolled.

Exclusion Criteria:

* Subjects who cannot understand the Italian language and who do not provide consent to study will be excluded.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 79 (Actual)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-05-15 (Actual)

PRIMARY OUTCOMES:
intensity of pain | The pain will be detected 3 times a day (8am/2 pm/8 pm) starting from the day of the first rehabilitation treatment until the fifth postoperative day.
  numeric rating scale (NRS) (from 0 to 10); The 11-point numerical scale ranges from "0" representing one pain extreme (eg "No pain") to "10" representing the other pain extreme (eg "More severe pain than you can imagine" or "worst pain imaginable").

SECONDARY OUTCOMES:
intensity of pain (short term) | the values of the NRS scale will be detected before and after the rehabilitation treatment up to fifth day
  numeric rating scale (NRS) (from 0 to 10); The 11-point numerical scale ranges from "0" representing one pain extreme (eg "No pain") to "10" representing the other pain extreme (eg "More severe pain than you can imagine" or "worst pain imaginable").
TUG - Time Up and Go | the TUG test will be administered during the 5th postoperative day
  Timed up and go is a simple test to measure a person's mobility level and requires static and dynamic balancing skills. It consists of measuring how many seconds it takes the patient to get up from the chair, walk a distance of 3 meters, turn around, return to the chair and sit down again.

CONTACTS AND LOCATIONS:
Overall Officials: antonio culcasi, PT, Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lotan S, Kalichman L. Manual therapy treatment for adolescent idiopathic scoliosis. J Bodyw Mov Ther. 2019 Jan;23(1):189-193. doi: 10.1016/j.jbmt.2018.01.005. Epub 2018 Feb 3. PMID 30691751
- [Background] Agabegi SS, Kazemi N, Sturm PF, Mehlman CT. Natural History of Adolescent Idiopathic Scoliosis in Skeletally Mature Patients: A Critical Review. J Am Acad Orthop Surg. 2015 Dec;23(12):714-23. doi: 10.5435/JAAOS-D-14-00037. Epub 2015 Oct 28. PMID 26510624
- [Background] Lamontagne LL, Hepworth JT, Salisbury MH. Anxiety and postoperative pain in children who undergo major orthopedic surgery. Appl Nurs Res. 2001 Aug;14(3):119-24. doi: 10.1053/apnr.2001.24410. PMID 11481590
- [Background] Sjoling M, Nordahl G, Olofsson N, Asplund K. The impact of preoperative information on state anxiety, postoperative pain and satisfaction with pain management. Patient Educ Couns. 2003 Oct;51(2):169-76. doi: 10.1016/s0738-3991(02)00191-x. PMID 14572947
- [Background] Ballantyne JC, Carr DB, deFerranti S, Suarez T, Lau J, Chalmers TC, Angelillo IF, Mosteller F. The comparative effects of postoperative analgesic therapies on pulmonary outcome: cumulative meta-analyses of randomized, controlled trials. Anesth Analg. 1998 Mar;86(3):598-612. doi: 10.1097/00000539-199803000-00032. PMID 9495424
- [Background] Joshi GP, Ogunnaike BO. Consequences of inadequate postoperative pain relief and chronic persistent postoperative pain. Anesthesiol Clin North Am. 2005 Mar;23(1):21-36. doi: 10.1016/j.atc.2004.11.013. PMID 15763409
- [Background] Beaulieu P, Cyrenne L, Mathews S, Villeneuve E, Vischoff D. Patient-controlled analgesia after spinal fusion for idiopathic scoliosis. Int Orthop. 1996;20(5):295-9. doi: 10.1007/s002640050081. PMID 8930721
- [Background] Vitale MG, Choe JC, Hwang MW, Bauer RM, Hyman JE, Lee FY, Roye DP Jr. Use of ketorolac tromethamine in children undergoing scoliosis surgery. an analysis of complications. Spine J. 2003 Jan-Feb;3(1):55-62. doi: 10.1016/s1529-9430(02)00446-1. PMID 14589246
- [Background] Wong GT, Yuen VM, Chow BF, Irwin MG. Persistent pain in patients following scoliosis surgery. Eur Spine J. 2007 Oct;16(10):1551-6. doi: 10.1007/s00586-007-0361-7. Epub 2007 Apr 5. PMID 17410382
- [Background] Kotzer AM. Factors predicting postoperative pain in children and adolescents following spine fusion. Issues Compr Pediatr Nurs. 2000 Apr-Jun;23(2):83-102. doi: 10.1080/01460860050121411. PMID 11111499
- [Background] Busch V, Magerl W, Kern U, Haas J, Hajak G, Eichhammer P. The effect of deep and slow breathing on pain perception, autonomic activity, and mood processing--an experimental study. Pain Med. 2012 Feb;13(2):215-28. doi: 10.1111/j.1526-4637.2011.01243.x. Epub 2011 Sep 21. PMID 21939499
- [Background] Janssens L, Brumagne S, McConnell AK, Hermans G, Troosters T, Gayan-Ramirez G. Greater diaphragm fatigability in individuals with recurrent low back pain. Respir Physiol Neurobiol. 2013 Aug 15;188(2):119-23. doi: 10.1016/j.resp.2013.05.028. Epub 2013 May 31. PMID 23727158
- [Background] Bordoni B, Marelli F. Failed back surgery syndrome: review and new hypotheses. J Pain Res. 2016 Jan 12;9:17-22. doi: 10.2147/JPR.S96754. eCollection 2016. PMID 26834497
- [Background] Kolar P, Sulc J, Kyncl M, Sanda J, Cakrt O, Andel R, Kumagai K, Kobesova A. Postural function of the diaphragm in persons with and without chronic low back pain. J Orthop Sports Phys Ther. 2012 Apr;42(4):352-62. doi: 10.2519/jospt.2012.3830. Epub 2011 Dec 21. PMID 22236541
- [Background] Marti-Salvador M, Hidalgo-Moreno L, Domenech-Fernandez J, Lison JF, Arguisuelas MD. Osteopathic Manipulative Treatment Including Specific Diaphragm Techniques Improves Pain and Disability in Chronic Nonspecific Low Back Pain: A Randomized Trial. Arch Phys Med Rehabil. 2018 Sep;99(9):1720-1729. doi: 10.1016/j.apmr.2018.04.022. Epub 2018 May 19. PMID 29787734
- [Background] Grams ST, Ono LM, Noronha MA, Schivinski CI, Paulin E. Breathing exercises in upper abdominal surgery: a systematic review and meta-analysis. Rev Bras Fisioter. 2012 Sep-Oct;16(5):345-53. doi: 10.1590/s1413-35552012005000052. Epub 2012 Oct 9. PMID 23060237
- [Background] Cloyd C, Moffett BS, Bernhardt MB, Monico EM, Patel N, Hanson D. Efficacy of liposomal bupivacaine in pediatric patients undergoing spine surgery. Paediatr Anaesth. 2018 Nov;28(11):982-986. doi: 10.1111/pan.13482. Epub 2018 Sep 11. PMID 30207019
- [Background] Covotta M, Claroni C, Costantini M, Torregiani G, Pelagalli L, Zinilli A, Forastiere E. The Effects of Ultrasound-Guided Transversus Abdominis Plane Block on Acute and Chronic Postsurgical Pain After Robotic Partial Nephrectomy: A Prospective Randomized Clinical Trial. Pain Med. 2020 Feb 1;21(2):378-386. doi: 10.1093/pm/pnz214. PMID 31504875
- [Background] Delage N, Morel V, Picard P, Marcaillou F, Pereira B, Pickering G. Effect of ketamine combined with magnesium sulfate in neuropathic pain patients (KETAPAIN): study protocol for a randomized controlled trial. Trials. 2017 Nov 3;18(1):517. doi: 10.1186/s13063-017-2254-3. PMID 29100524
- [Background] Stienen MN, Maldaner N, Joswig H, Corniola MV, Bellut D, Prommel P, Regli L, Weyerbrock A, Schaller K, Gautschi OP. Objective functional assessment using the "Timed Up and Go" test in patients with lumbar spinal stenosis. Neurosurg Focus. 2019 May 1;46(5):E4. doi: 10.3171/2019.2.FOCUS18618. PMID 31042663
- [Background] Gautschi OP, Joswig H, Corniola MV, Smoll NR, Schaller K, Hildebrandt G, Stienen MN. Pre- and postoperative correlation of patient-reported outcome measures with standardized Timed Up and Go (TUG) test results in lumbar degenerative disc disease. Acta Neurochir (Wien). 2016 Oct;158(10):1875-81. doi: 10.1007/s00701-016-2899-9. Epub 2016 Aug 3. PMID 27488842
- [Background] Ross MC, Bohannon AS, Davis DC, Gurchiek L. The effects of a short-term exercise program on movement, pain, and mood in the elderly. Results of a pilot study. J Holist Nurs. 1999 Jun;17(2):139-47. doi: 10.1177/089801019901700203. PMID 10633648
- [Background] Anderson BE, Bliven KCH. The Use of Breathing Exercises in the Treatment of Chronic, Nonspecific Low Back Pain. J Sport Rehabil. 2017 Sep;26(5):452-458. doi: 10.1123/jsr.2015-0199. Epub 2016 Aug 24. PMID 27632818
- [Background] Jafari H, Courtois I, Van den Bergh O, Vlaeyen JWS, Van Diest I. Pain and respiration: a systematic review. Pain. 2017 Jun;158(6):995-1006. doi: 10.1097/j.pain.0000000000000865. PMID 28240995
- [Background] Sloman R, Wruble AW, Rosen G, Rom M. Determination of clinically meaningful levels of pain reduction in patients experiencing acute postoperative pain. Pain Manag Nurs. 2006 Dec;7(4):153-8. doi: 10.1016/j.pmn.2006.09.001. PMID 17145489
- [Background] Rakel B, Herr K. Assessment and treatment of postoperative pain in older adults. J Perianesth Nurs. 2004 Jun;19(3):194-208. doi: 10.1016/j.jopan.2004.03.005. PMID 15195278